CLINICAL TRIAL: NCT02121223
Title: A Prospective, Multi-center,Randomized Controled Trial of POST-dilatation to Improve Outcomes in Acute STEMI Patients Undergoing Primary PCI After Thrombus Aspiration and DES Implantation With OCT Assessment
Brief Title: POST-dilatation to Improve Outcomes in Acute STEMI Patients Undergoing Primary With OCT Assessment
Acronym: POST-STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai East Hospital (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, Professor, Chief of Heart Center, and President of the Hospital, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZJU CT002
Record Dates: First submitted 2014-04-03; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Acute Myocardial Infarction
Keywords: acute ST segment elevated myocardial infarction; primary percutaneous intervention; Stent Incomplete Apposition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Patients in control group will receive current standard therapy for STEMI: manual thrombus aspiration + Promus Element stent implantation ( with a pressure less than 12 atm), but not post-dilatation
  Interventions: Device: manual thrombus aspiration + Promus Element stent implant
- Post-dilatation (Experimental): Patients in this group will receive high pressure post-dilatation with a Quantum Maverick balloon after manual thrombus aspiration + Promus Element stent implantation
  Interventions: Device: post-dilatation with a Quantum Maverick balloon; Device: manual thrombus aspiration + Promus Element stent implant

INTERVENTIONS:
Device: post-dilatation with a Quantum Maverick balloon — post-dilatation with a Quantum Maverick balloon at high pressure (>=16atm) for at least 15 seconds.
  Arms: Post-dilatation
Device: manual thrombus aspiration + Promus Element stent implant — manual thrombus aspiration followed by Promus Element stent implantation at normal pressure

SUMMARY:
To evaluate the effective and safety of post-dilatation in patients with acute ST segment elevated myocardial infarction undergoing primary percutaneous intervention after thrombus aspiration assessed by optical coherence tomography to examine stent Incomplete apposition and strut coverage in patients treated with drug-eluting stents .

ELIGIBILITY:
Clinical Inclusion Criteria:

* Age ≥18 years
* STEMI >20 mins and <12 hours in duration
* ST-segment elevation of ≥1 mm in ≥2 contiguous leads; or Presumably new left bundle branch block; or True posterior MI with ST depression of ≥1 mm in ≥2 contiguous anterior leads
* Written, informed consent

Angiographic Inclusion Criteria

* The presence of least 1 acute infarct artery target vessel* in which:

  1. ALL significant lesions are eligible for stenting with study stents, and
  2. ALL such lesions have a visually estimated reference diameter ≥2.5 mm and ≤4.0 mm
  3. All culprit lesion TIMI Flow ≤ 0 or 1 Grade prior to guide wire crossing
* Expected ability to deliver the stent(s) to all culprit lesions (absence of excessive proximal tortuosity or severe calcification)
* Expected ability to fully expand the stent(s) at all culprit lesions (absence of marked calcification)

Clinical Exclusion Criteria:

* Contraindication to any of the study medications
* Patients with cardiogenic shock
* History of bleeding diathesis or known coagulopathy , or will refuse blood transfusions
* History of intracerebral mass, aneurysm, AVM, or hemorrhagic stroke; stroke or TIA within 6 months or any permanent neurologic deficit; GI or GU bleed within 2 months, or major surgery within 6 weeks; recent or known platelet count <100,000 cells/mm3 or hgb <10 g/dL
* Planned elective surgical procedure that would necessitate interruption of thienopyridines during the first 6 months post enrollment

Angiographic Exclusion Criteria

* Bifurcation lesion definitely requiring implantation of stents in both the main vessel + side branch
* Infarct related artery is an unprotected left main
* >38 mm of study stent length anticipated
* Infarction due to stent thrombosis, or infarct lesion at the site of a previously implanted stent
* High likelihood of CABG within 30 days anticipated
* The culprit lesion will be judged unsuitable for OCT procedure, because of conditions such as left main trunk disease or shock vital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Incomplete Stent Apposition (ISA) in OCT at 7 month | 7 months after primary PCI

SECONDARY OUTCOMES:
Final TIMI flow grade 3 | Immediately after primary PCI procedure (up to 2 min)
Final TIMI blush Grade 3 | Immediately after primary PCI procedure (up to 2 min)
Rate of ST resolution 70% at 30 day | 30 days after primary PCI
Rate of strut coverage in OCT at 7 month | 7 months after primary PCI
MACE at 7 month and 12 month | 7 months and 12 months after primary PCI
TLR ,TLF at 7 month and 12 month | 7 months and 12months after primary PCI
Stent thrombus rate at 30 day,7 month and 12 month | 30 days, 7 months and 12 months after primary PCI
In-stent and in-segment late loss | 7 months after primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Jiang J, Tian NL, Cui HB, Li CL, Liu XB, Dong L, Sun Y, Chen XM, Chen SL, Xu B, Wang JA. Post-dilatation improves stent apposition in patients with ST-segment elevation myocardial infarction receiving primary percutaneous intervention: A multicenter, randomized controlled trial using optical coherence tomography. World J Emerg Med. 2020;11(2):87-92. doi: 10.5847/wjem.j.1920-8642.2020.02.004. PMID 32076473